CLINICAL TRIAL: NCT05148741
Title: Evaluation of Capsular Bag Shape Changes After Plate-haptic Intraocular Lens Implantation by SS-OCT.
Status: Completed | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Other Study IDs: SS-OCT plate-haptic
Record Dates: First submitted 2021-09-14; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Age-related Cataract
Keywords: SS-OCT; capsule bag

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: implanted with the C-loop haptic intraocular lens
- Group 2: implanted with the plate haptic intraocular lens

SUMMARY:
Evaluation of capsular bag shape changes after plate-haptic intraocular lens implantation by SS-OCT.

DETAILED DESCRIPTION:
Eighty patients (80 eyes) with simple age-related cataracts were treated from December 2019 to December 2020 in the Wenzhou Medical University. Investigators specifically included patients who were bodily healthy and underwent a successful implantation of an IOL. Inclusion criteria for this study were patients who were older than 40 years old, had an axial length of 22-26mm, and could complete 4 follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

-patients who were older than 40 years old, had an axial length of 22-26mm, and could complete 4 follow-up visits.

Exclusion Criteria:

* people cannot cooperate with the check， corneal opacity, glaucoma, and other eye diseases
* any other previous intraocular surgery, and intraoperative complications including anterior or posterior capsulartears
* Continuous circular capsulorhexis is not centered and Mydriasis is less than 7mm.

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients were divided into 2 groups according to the different intraocular lenses implanted: 39 eyes were implanted with the C-loop haptic intraocular lens (Acrysof) while the other 41 eyes were implanted with plate haptic intraocular lenses (CT ASPHINA 509 M).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Capsular bend index (CBI) | 2020.12.1
  capsule bend formation has 5 continuous stages from 0 to 4，The stage score varies over different positions of the same capsule bag, because the capsule bend formation is inconsistent along the entire optic edge. CBI is the mean of the different stage scores in different positions and represents the general capsule bend state of the whole capsule bag.

CONTACTS AND LOCATIONS:
Overall Officials: Yune Zhao, Study Director — Ophthalmology and Optometry Hospital
Locations (1):
- Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China